CLINICAL TRIAL: NCT02278666
Title: Minimally Invasive Aortic Valve Replacement Versus Conventional Aortic Valve Replacement: a Long Term Registry on Potential Benefits of the Different Surgical Techniques
Brief Title: Minimally Invasive Versus Conventional Aortic Valve Replacement: a Long Term Registry
Acronym: SATURNO
Status: Completed | Type: Observational
Sponsor: Maria Cecilia Hospital (Other)
Collaborators: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESREFO21
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2022-07

CONDITIONS: Aortic Valve Surgery
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- upper mini-sternotomy: aortic valve replacement surgery via upper J or T sternotomy (ministernotomy)
  Interventions: Procedure: aortic valve replacement; Device: biological prosthetic valve; Device: Mechanical valve
- right mini thoracotomy: aortic valve replacement/repair surgery via right mini thoracotomy
  Interventions: Procedure: aortic valve replacement; Device: biological prosthetic valve; Device: Mechanical valve
- conventional sternotomy: aortic valve replacement surgery via conventional full sternotomy
  Interventions: Procedure: aortic valve replacement; Device: biological prosthetic valve; Device: Mechanical valve

INTERVENTIONS:
Procedure: aortic valve replacement — aortic valve replacement with either biological prosthetic valve or mechanical valve
  Other Names: AVR
Device: biological prosthetic valve — aortic valve replacement with either biological prosthetic valve or mechanical valve
Device: Mechanical valve — aortic valve replacement with either biological prosthetic valve or mechanical valve

SUMMARY:
The aim of the present study is to assess in a "real life" case list the outcome of three different surgical approaches for isolated aortic valve surgery in terms of surgery times, morbidity and mortality.

DETAILED DESCRIPTION:
The study will focus on data recorded and collected from daily clinical treatment of patients undergoing isolated aortic valve replacement due to symptomatic aortic stenosis who consented to the use of their personal data. After surgery patients will be followed up to a minimum of 12 months. In-hospital and follow-up outcomes of the different surgical approaches will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing isolated aortic valve surgery
* Written Informed consent to the use of personal data

Exclusion Criteria:

* other associated cardiac surgery
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing isolated aortic valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary bypass time | during surgery
Total duration of Intensive Care Unit stay | during hospital stay, usually lasting one to two weeks
Blood transfusions | during hospital stay, usually lasting one to two weeks

SECONDARY OUTCOMES:
renal insufficiency | during hospital stay, usually lasting one to two weeks
  need for haemofiltration
Prolonged ventilation | during hospital stay
  longer than 24 hours
Re-exploration for bleeding | during hospital stay, usually lasting one to two weeks
  need of surgical revision for bleeding
sepsis | during hospital stay, usually lasting one to two weeks
Neurological complications | during hospital stay, usually lasting one to two weeks
  stroke and/or transient ischemic attacks
in-hospital mortality | during hospital stay, usually lasting one to two weeks
30-day mortality | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mikus, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy